CLINICAL TRIAL: NCT04884672
Title: Post-Market Clinical Follow-up Study on SMILE Treatment of Myopia With and Without Astigmatism by VISUMAX 800
Brief Title: PMCF Study on SMILE Treatment of Myopia With and Without Astigmatism
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Collaborators: In Vitro Research Solutions Pvt Ltd (iVRS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: V1902PM
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Myopia; Astigmatism
Keywords: SMILE; Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SMILE — Small incision lenticule extraction, a refractive surgery procedure for the corrcetion of myopia with or without astigmatism

SUMMARY:
The primary objective of this PMCF investigation is to systematically collect safety and effectiveness data with the VISUMAX 800 laser in clinical daily routine SMILE use for the purpose of post market surveillance.

DETAILED DESCRIPTION:
The present PMCF study is a prospective, non-randomized, international multi-center study without control group including patients with myopia or myopia combined with astigmatism undergoing SMILE with the VISUMAX 800 femtosecond laser in daily routine use.

In this PMCF study, at maximum 474 eyes of consecutive subjects will be consented, enrolled, treated and followed up to 6 months postoperatively at 4 to 5 sites. The treatments, which will be done bilateral, shall be equally distributed between the sites as far as possible.

The subjects will be 18 years of age or older, who suffer from myopia of up to -10 D with or without astigmatism of up to 5 D, and are suitable for SMILE treatments, fulfil all inclusion criteria and not fulfil any of the exclusion criteria.

The expected duration of the is 16 months (site initiation to closeout visit).

ELIGIBILITY:
Inclusion Criteria:

* Myopia up to -10 D with and without astigmatism up to 5 D
* Age of 18 years or older
* Pre-operative CDVA of 20/25 or better in each eye
* Patient shall be willing to comply with all follow-up visits and the respective examinations
* Patients should be able to understand the patient information and willing to sign an informed consent.
* Contact lens wearers must stop wearing their contact lenses at least 2 weeks before baseline measurements in case of hard contact lenses and 2 days before baseline measurements in case of soft contact lenses

Exclusion Criteria:

* No monovision treatments (target sphere may not be more negative than -0.25 D)
* The patient may not participate in other ophthalmologic studies except in VEMOS study at site Aarhus.
* Any impaired person (minors, pregnant or breast-feeding women or persons incapable of giving consent) are definitely excluded from the study.
* The patients presenting at least one of the contraindications stated in User Manual of the VISUMAX 800 option ReLEx SMILE must not be included in this clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the device are patients with myopia and myopia combined with astigmatism, who are medically suitable for femtosecond laser treatment with the SMILE treatment.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Accuracy of manifest spherical equivalent | 1 week
  Determination of the percentage of eyes with MRSE-target SE within
  ±0.5D with a half width of 95% confidence-interval of 4%
Accuracy of manifest spherical equivalent | 1 month
  Determination of the percentage of eyes with MRSE-target SE within
  ±0.5D with a half width of 95% confidence-interval of 4%
Accuracy of manifest spherical equivalent | 3 months
  Determination of the percentage of eyes with MRSE-target SE within
  ±0.5D with a half width of 95% confidence-interval of 4%
Accuracy of manifest spherical equivalent | 6 months
  Determination of the percentage of eyes with MRSE-target SE within
  ±0.5D with a half width of 95% confidence-interval of 4%
Accuracy of astigmatism | 1 week
  Determination of the percentage of eyes with absolute post-OP astigmatism within ±0.5D with a half width of 95% confidence-interval of 4%
Accuracy of astigmatism | 1 month
  Determination of the percentage of eyes with absolute post-OP astigmatism within ±0.5D with a half width of 95% confidence-interval of 4%
Accuracy of astigmatism | 3 months
  Determination of the percentage of eyes with absolute post-OP astigmatism within ±0.5D with a half width of 95% confidence-interval of 4%
Accuracy of astigmatism | 6 months
  Determination of the percentage of eyes with absolute post-OP astigmatism within ±0.5D with a half width of 95% confidence-interval of 4%
Early visual acuity | 1 day
  Determination of the difference between post-operative UDVA and pre-operative CDVA with a half width of 95% confidence-interval of 0.02 logMAR
Early visual acuity | 1 week
  Determination of the difference between post-operative UDVA and pre-operative CDVA with a half width of 95% confidence-interval of 0.02 logMAR
Side effects and complications | 1 day
  Determination of the rates of side effects and intra-operative complications with an accuracy, which in case of a zero frequency allows the conclusion of being lower or equal than 1%, which means that the upper confidence limit is 1%.
Side effects and complications | 1 week
  Determination of the rates of side effects and intra-operative complications with an accuracy, which in case of a zero frequency allows the conclusion of being lower or equal than 1%, which means that the upper confidence limit is 1%.
Side effects and complications | 1 month
  Determination of the rates of side effects and intra-operative complications with an accuracy, which in case of a zero frequency allows the conclusion of being lower or equal than 1%, which means that the upper confidence limit is 1%.
Side effects and complications | 3 months
  Determination of the rates of side effects and intra-operative complications with an accuracy, which in case of a zero frequency allows the conclusion of being lower or equal than 1%, which means that the upper confidence limit is 1%.
Side effects and complications | 6 months
  Determination of the rates of side effects and intra-operative complications with an accuracy, which in case of a zero frequency allows the conclusion of being lower or equal than 1%, which means that the upper confidence limit is 1%.

SECONDARY OUTCOMES:
CDVA | 1 week
  Distribution of post-op CDVA change against baseline and Cumulative distribution of post-operative CDVA
CDVA | 1 month
  Distribution of post-op CDVA change against baseline and Cumulative distribution of post-operative CDVA
CDVA | 3 months
  Distribution of post-op CDVA change against baseline and Cumulative distribution of post-operative CDVA
CDVA | 6 months
  Distribution of post-op CDVA change against baseline and Cumulative distribution of post-operative CDVA
Mesopic contrast sensitivity | 6 months
  Mesopic contrast sensitivity and change against baseline
UDVA | 1 day
  Cumulative distribution of post-op UDVA (compared to pre-op CDVA) and Distribution of change of UDVA against pre-op CDVA (in units of lines)
UDVA | 1 week
  Cumulative distribution of post-op UDVA (compared to pre-op CDVA) and Distribution of change of UDVA against pre-op CDVA (in units of lines)
UDVA | 1 month
  Cumulative distribution of post-op UDVA (compared to pre-op CDVA) and Distribution of change of UDVA against pre-op CDVA (in units of lines)
UDVA | 3 months
  Cumulative distribution of post-op UDVA (compared to pre-op CDVA) and Distribution of change of UDVA against pre-op CDVA (in units of lines)
UDVA | 6 months
  Cumulative distribution of post-op UDVA (compared to pre-op CDVA) and Distribution of change of UDVA against pre-op CDVA (in units of lines)
Predictability and accuracy | 1 week
  Predictability plots for attempted versus achieved MRSE including regression analysis and Predictability of astigmatism (vector based) including regression analysis. and Accuracy plots (distribution of pre and post-op MRSE and Astigmatim) and Induced astigmatism
Predictability and accuracy | 1 month
  Predictability plots for attempted versus achieved MRSE including regression analysis and Predictability of astigmatism (vector based) including regression analysis. and Accuracy plots (distribution of pre and post-op MRSE and Astigmatim) and Induced astigmatism
Predictability and accuracy | 3 months
  Predictability plots for attempted versus achieved MRSE including regression analysis and Predictability of astigmatism (vector based) including regression analysis. and Accuracy plots (distribution of pre and post-op MRSE and Astigmatim) and Induced astigmatism
Predictability and accuracy | 6 months
  Predictability plots for attempted versus achieved MRSE including regression analysis and Predictability of astigmatism (vector based) including regression analysis. and Accuracy plots (distribution of pre and post-op MRSE and Astigmatim) and Induced astigmatism
Stability | between 1 month 3 months
  Stability of MRSE and Astigmatism (change between 2 consecutive timepoints)
Stability | between 3 months and 6 months
  Stability of MRSE and Astigmatism (change between 2 consecutive timepoints)
Cylinder vector analyses | 1 week
  Cylinder vector analyses as double angle plots as well as descriptive statistics on:
  target induced astigmatism, surgical induced astigmatism, correction index, index of success, angle of error, magnitude of error.
Cylinder vector analyses | 1 month
  Cylinder vector analyses as double angle plots as well as descriptive statistics on:
  target induced astigmatism, surgical induced astigmatism, correction index, index of success, angle of error, magnitude of error.
Cylinder vector analyses | 3 months
  Cylinder vector analyses as double angle plots as well as descriptive statistics on:
  target induced astigmatism, surgical induced astigmatism, correction index, index of success, angle of error, magnitude of error.
Cylinder vector analyses | 6 months
  Cylinder vector analyses as double angle plots as well as descriptive statistics on:
  target induced astigmatism, surgical induced astigmatism, correction index, index of success, angle of error, magnitude of error.
Patient Questionnaire | 6 months
  Aspects of PROWL patient questionnaire. Change against baseline.
Corneal wave-front, change against baseline | 6 months
  Simple statistics on corneal wave-front parameters (higher order RMS, Coma and Spherical aberration)
Centration | during the procedure
  Analysis of achieved centration based on centration parameters of device.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Hjortdal, Prof., Principal Investigator — Department of Clinical Medicine - Department of Ophthalmology
Locations (5):
- Department of Clinical Medicine - Department of Ophthalmology, Aarhus, Denmark
- Germany (2):
  - University Medical Center Universitätsklinikum Gießen Marburg, Marburg
  - Smile Eyes Airport München, München
- HKSH Healthcare Guy Hugh Chan Refractive Surgery Centre, Hong Kong, Hong Kong
- Medical Center Nethradhama Superspeciality Eye Hospital, Bangalore, India

IPD SHARING:
Plan to Share IPD: No
There is no data sharing planned.